CLINICAL TRIAL: NCT06630936
Title: Prospective Multi-Center Cohort Study of Atrial Fibrillation Combined with Atrial Functional Mitral Regurgitation
Brief Title: Study of Atrial Fibrillation Combined with Atrial Functional Mitral Regurgitation
Acronym: AFMR
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0882
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation (AF); Atrial Functional Mitral Regurgitation
Keywords: Atrial Fibrillation; Atrial Functional Mitral Regurgitation; catheter ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Catheter ablation cohort: Patients who receive pulsed field ablation procedure
- Drug treatment cohort: Patients who receive regular drug therapy

SUMMARY:
To evaluate the improvement of mitral regurgitation after catheter ablation of atrial fibrillation or regular drug therapy in atrial fibrillation patients combined with atrial functional mitral regurgitation.

DETAILED DESCRIPTION:
Atrial fibrillation results in the loss of the atria's normal contracting ability, leading to blood stasis within the left atrium and its subsequent enlargement. This condition can progress to cause dilation of the mitral annulus and mitral regurgitation-a phenomenon referred to as functional mitral regurgitation (FMR). Atrial functional mitral regurgitation (AFMR), triggered by the enlargement of the left atrium and remodeling of the mitral annulus, has increasingly become a focal point of research in recent times. Past studies have indicated that in patients who revert to and maintain sinus rhythm following catheter ablation for atrial fibrillation, there is a notable reduction in the size of the left atrium, the diameter of the mitral annulus, and the severity of mitral regurgitation. This suggests that patients with AFMR may derive significant benefits from the restoration of sinus rhythm. This investigation constitutes a prospective, multicenter cohort study. Eligible patients diagnosed with atrial fibrillation accompanied by atrial functional mitral regurgitation, who meet the inclusion criteria and do not fulfill the exclusion criteria, are being recruited. Depending on clinical judgment or patient preference, participants are assigned to receive either catheter ablation for atrial fibrillation or standard medical therapy, with the aim of assessing the impact of these different treatments on alleviating the degree of mitral regurgitation. The study aims to enroll 500 patients, with follow-up assessments scheduled at 3-month, 6-month, and 12-month intervals following enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years old;
2. Patients diagnosed with symptomatic paroxysmal atrial fibrillation (AF history < 5 years)
3. Moderate to severe MR and normal LV ejection fraction (≥50%), LVEDD<55 mm, and normal LV wall systolic function
4. Able to understand the purpose of the trial, participate in the trial voluntarily with informed consent form signed by the subject him/herself or his or her legal representative, and willing to complete follow-up visits as required under the protocol

Exclusion Criteria:

1. Atrial fibrillation secondary to electrolyte imbalances, thyroid disease or other reversible factors
2. Active endocarditis or active rheumatic heart disease, or degenerative mitral regurgitation due to endocarditis or rheumatic valvular heart disease
3. Moderate to severe mitral stenosis
4. Imaging examination shows left atrium or left atrial appendage thrombosis
5. Left ventricular ejection fraction less than 50%
6. Left atrial diameter more than 50mm
7. Patients with previous left atrial appendage occlusion or left atrial appendage closure, patent foramen ovale closure, atrial septal defect closure or repair (only applied for patients who need to ablation)
8. Patients who have implanted devices such as implantable cardioverter defibrillator(ICD), cardiac resynchronization therapy(CRT) or pacemaker
9. Previous metal artificial valve or valve repair device implantation (only applied for patients who need to ablation)
10. Presence of lateral thrombus, tumors or other abnormalities that interfere with vascular puncture or catheter operation (only applied for patients who need to ablation)
11. Anticoagulation contraindications, and history of blood clotting or bleeding abnormalities
12. Acute systemic infection
13. Female patients who are pregnant, lactating, or unable to use contraception during the study
14. Patients' life expectancy is less than 12 months
15. Abnormalities or diseases that the investigator believes should be excluded from the scope of enrollment in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation combined with atrial functional mitral regurgitation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement in MR | 3-month, 6-month, 12-month at follow-up
  Defined as a decrease of ≥1 level in the severity stage at 1 year compared to baseline

SECONDARY OUTCOMES:
Changes of MR in echocardiography examination | 3-month, 6-month, 12-month at follow-up
  Effective regurgitant area, regurgitant volume, and regurgitant fraction of the mitral valve from baseline
Changes of left ventricular function in echocardiography examination | 3-month, 6-month, 12-month at follow-up
  Left ventricular ejection fraction, end-systolic/end-diastolic volume, end-systolic/end-diastolic diameter, early diastolic mitral valve flow velocity E, mitral annular velocity e'at the septum and lateral wall, and E/e'
Changes of left atrial function in echocardiography examination | 3-month, 6-month, 12-month at follow-up
  Left atrial anteroposterior diameter and left atrial end-diastolic volume
Freedom from atrial arrhythmia recurrence | 12-month at follow-up
  Defined as ECG data (including surface ECG and 24-h Holter) during the efficacy evaluation period (blanking period to the end of the 12-month follow-up) without recording AF, AFL, or AT (arrhythmia monitoring device ≥ 30 s)
Burden of atrial arrhythmia | 12-month at follow-up
  Incidence and duration of atrial arrhythmias (atrial premature contractions, atrial tachycardia, atrial flutter, and atrial fibrillation)
Acute PVI success | Immediately after cathete ablation procedure
  Immediate success rate of pulmonary vein isolation
Procedure time | Immediately after cathete ablation procedure
  Total procedure time, atrial fibrillation ablation time, radiofrequency energy time, and total fluoroscopy time
Incidence rate of major adverse events | 3-month, 6-month, 12-month at follow-up
  death, myocardial infarction, pulmonary vein stenosis, diaphragmatic nerve palsy, systemic embolism, TIA/ischemic stroke, pericarditis, pericardial effusion/cardiac tamponade, atrioesophageal fistula, and severe vascular access complications
Incidence of heart failure-related events | 3-month, 6-month, 12-month at follow-up
  Including readmissions, stroke, and all-cause mortality
Changes in QoL | 3-month, 6-month, 12-month at follow-up
  KCCQ score and NYHA classification

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, Dorctor, Principal Investigator — Second Affiliated Hospital of Zhejiang University, School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No